CLINICAL TRIAL: NCT04051970
Title: Randomized, Open-label, Phase III Trial Comparing a Dual Nucleoside Analogues Strategy Preceded by a Triple Therapy Induction Period to an Immediate Strategy With Dolutegravir Plus Lamivudine in Antiretriviral naïve People Living With HIV With Viral Load < 50000 cp/mL and CD4 Cells >300/mm3
Brief Title: Reducing Antiretroviral Treatments
Acronym: ALTAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 173
Record Dates: First submitted 2019-07-26; First posted 2019-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Anti-Retroviral Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy TRI-BI (Experimental)
  Interventions: Drug: Antiretroviral
- Strategy Immediate BI (Active Comparator)
  Interventions: Drug: Antiretroviral

INTERVENTIONS:
Drug: Antiretroviral — Antiretroviral treatments (ART) will be allocated through central randomization (1:1:) according to the following two strategies:
  Tritherapy-Bitherapy (TRI-BI) strategy:
  TRI between D0 and W16: 3-drug combination (3-DR) including 2 NRTI (either TDF or TAF+XTC) and a once daily integrase inhibitor (Stribild® or Genvoya® or Biktarvy®) or TDF/XTC Gé + Tivicay® or TDF/XTC Gé + Isentress® QD 1200 mg when available) during 16 weeks BI between W16 and W96: if pVL viral load <500 cp/mL at W4 and <50 cp/mL at W12, participants will start the 2-DR regimen TDF or TAF / XTC (TDF/XTC Gé or Descovy®) at W16, until W96.
  (Descovy® : provided that it is available in France), (XTC = FTC or 3TC)
  Immediate Bitherapy (BI) strategy Dolutegravir (DTG, Tivicay® 50 mg QD) plus lamivudine (3TC, 300 mg QD) between D0 and W96.
  Antiretroviral drugs will be prescribed in the context of standard of care.

SUMMARY:
The purpose of this trial is to demonstrate at W48 the non-inferiority of a dual nucleoside analogues strategy with tenofovir (TDF) or tenofovir alafenamide (TAF) plus emtricitabine (FTC) or lamivudine (3TC) preceded by a 16 week induction period with TDF or TAF plus FTC or 3TC plus an integrase inhibitor (INI) relative to an immediate 2-DR strategy with dolutegravir plus 3TC in HIV-infected antiretroviral therapy (ARV) naïve participants with CD4 cells count greater than 300/mm3 and a low viral load defined as plasma HIV RNA strictly lower than 50 000 cp/mL

DETAILED DESCRIPTION:
ANRS 173 ALTAR is a multicenter, comparative, international, open label, phase III randomized trial aiming at evaluating the non-inferiority of a TRI-BI (tritherapy-bitherapy) strategy (includes a 16 week - induction phase with 2 NRTI and a once daily integrase inhibitor followed by a bitherapy with TDF or TAF / XTC*) in its capacity to achieve viral suppression at week 48 versus immediate BI (bitherapy) strategy (DTG/3TC) in participants naïve to antiretroviral therapy with plasma HIV RNA strictly less than 50 000 copies/mL and CD4 cells count above 300/mm3.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection (positive HIV-1 serology or plasma viral load)
* Age ≥ 18 years
* Therapeutic antiretroviral treatment-naive participant (history of prophylaxy is accepted)
* CD4 cells count > 300 cells/mm3 at screening visit
* HIV-1-RNA plasma viral load <50 000 copies/mL at screening visit
* Full susceptibility to trial drugs (NRTI, INI) at screening visit
* eGFR (epidermal growth factor receptor) > 60 mL /min (MDRD)
* AST (aspartate aminotransferase), ALT(alanine transaminase) < 3x norm
* Absence of any AIDS-defining event and/or opportunistic infection
* Possible contact by phone and/or email in order to be informed in case of detectable HIV plasma viral load
* Negative urinary pregnancy test at screening visit for women of childbearing age
* Written and informed consent signed
* For French participants only: subject enrolled in or a beneficiary of a Social Security programme (including State Medical Aid (AME), only if Ethic Committee approves it)

Exclusion Criteria:

* HIV-2 co-infection
* Hepatitis B Virus infection (positive HBs antigen)
* Any comorbidity potentially related to a life expectancy below 12 months
* Any condition (use of alcohol, drugs, etc.) judged by the investigator to possibly interfere with trial protocol compliance, adherence and/or trial treatment tolerance
* Pregnant women or breastfeeding women
* Women of childbearing age that do not want to use an effective method of contraception
* Participant under justice protection
* Galactose/lactose intolerance, Lapp lactase deficiency or glucose/galactose malabsorption (known or documented)
* Participation to another clinical trial evaluating a new treatment/therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate at W48 the non-inferiority | proportion of participants with plasma HIV-RNA <50 copies/mL at Week 48 in the 2 arms on allocated treatment (FDA snapshot approach)
  To demonstrate at W48 the non-inferiority of a dual nucleoside analogues strategy with tenofovir (TDF) or tenofovir alafenamide (TAF) plus emtricitabine (FTC) or lamivudine (3TC) preceded by a induction period with TDF or TAF plus FTC or 3TC plus an integrase inhibitor (INI) relative to an immediate 2-DR strategy with dolutegravir plus 3TC in HIV-infected ART naïve participants with CD4 cells count greater than 300/mm3 and a low viral load defined as plasma HIV RNA strictly lower than 50 000 cp/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital la Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No